CLINICAL TRIAL: NCT02389491
Title: Effect of a High Density Formula on Growth and Safety in Early Postoperative Infants With Congenital Heart Disease Duration of Cardiac Intensive Care Unit（CCU）Stay: a Randomized Clinical Trial
Brief Title: Effect of a High Density Formula on Growth and Safety in Congenital Heart Disease Infants
Acronym: CHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FNF201426
Record Dates: First submitted 2015-02-05; First posted 2015-03-17 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Congenital Heart Disease
Keywords: high density formula; heart defects; infant
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal density formula (Neocate) (Active Comparator): In control group,infants intake normal density formula (Neocate,67kcal/100ml) when starting enteral nutrition after operation and continue for 7days
  Interventions: Dietary Supplement: normal density formula (Necocate)
- high density formula (Infatrini) (Experimental): In the intervention group,infants intake high density formula (Infatrini, 100kcal/100ml) when starting enteral nutrition after operation and continue for 7days
  Interventions: Dietary Supplement: high density formula(Infatrini)

INTERVENTIONS:
Dietary Supplement: normal density formula (Necocate) — In control group,there are 32 infants
  Arms: normal density formula (Neocate)
Dietary Supplement: high density formula(Infatrini) — In intervention group,there are 32 infants
  Arms: high density formula (Infatrini)

SUMMARY:
The purpose of this study is to explore the effects of high density formula in early postoperative infants with congenital heart disease and to assess its safety.

DETAILED DESCRIPTION:
The number of infants born with CHD increases every year and most CHD infants are suffered with malnutrition.Recent studies have shown that increasing energy intake in CHD infants can improve their nutrition status.But there are no high qualified evidences supporting that high density formula can promote infants' nutrition status and ensure its safety. The hypothesis of the current study is that high density formula intake can increase infants'weight and it's safe.

The current study adopts randomized,controlled intervention trial, gives high density formula(Infatrini,100kcal/100ml)to CHD infants in intervention group and normal density formula（Neocate,67kcal/100ml）in control group. Intervention begins when infants start enteral nutrition after operation and continues for 7days.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of congenital heart disease from symptoms, signs, ultrasonic and imaging examination
2. aged from 1 day to 12 months
3. accept extracorporeal circulation open-heart surgery
4. family members voluntarily participate in this study

Exclusion Criteria:

1. patients have other diseases which cause nutrition disorders, such as gastrointestinal malformation, preoperative gastroesophageal reflux, genetic diseases related to the growth restriction
2. accept total parenteral nutrition
3. predicted the length of CCU stay is less than five days
4. patients have abdominal distention, diarrhea, vomiting

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
weight gain at the 7th day (g) | from the first day starting enteric feeding to the 7th days
  the 7th day body weight minus baseline body weight
the number of participants with feeding intolerance | from the first day starting enteric feeding to the 7th day
  Feeding intolerance means participants have gastric retention, vomiting, diarrhea ect. lead to enteric feeding was stopped.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  evaluate the long term effect of feeding high density formula
length of Cardiac Intensive Care Unit(CCU) stay | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  evaluate the long term effect of feeding high density formula
the number of participants with poor wound healing | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  evaluate the long term effect of feeding high density formula
the number of participants with necrotizing enterocolitis | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  evaluate the long term effect of feeding high density formula

CONTACTS AND LOCATIONS:
Overall Officials: Gu Ying, docter, Study Chair — Children Hospital of Fudan University